CLINICAL TRIAL: NCT06025006
Title: Impact of an Alternative to Incarceration by Housing and Support by Assertive Community Treatment Team (AILSI Program) for People Who Are Homeless With Severe Psychiatric Disorders and Referred to Referral Procedures, in Comparison With Usual Services: a Randomized Controlled Trial
Brief Title: Impact of an Alternative to Incarceration by Housing and Support by Assertive Community Treatment Team for Homeless People With Severe Psychiatric Disorders Referred to Referral Procedures : AILSI Program
Acronym: AILSI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-61
Record Dates: First submitted 2019-07-11; First posted 2023-09-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Severe Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AILSI (Experimental)
  Interventions: Other: alternative to incarceration
- the standard of care (No Intervention)

INTERVENTIONS:
Other: alternative to incarceration — place of respite with housing plus intensive follow-up
  Arms: AILSI

SUMMARY:
People who are homeless with severe psychiatric disorders have to negotiate discontinuous mental health care pathways including high use of emergency departement and enforced hospitalisation, poor access to ambulatory care, poor access to common rights services and a greater risk of incarceration.

In order to reduce morbidity, improve social integration and outpatient care for people with severe psychiatric disorders and multiple factors of social vulnerability, the concept of therapeutic jurisprudence has led to the emergence of mental health courts in Anglo-Saxon nations. These courts aim to condition alternatives to incarceration through community-based intensive care (assertive community treatment-ACT). ACT Teams offer direct access to housing without any prerequisite of treatment or abstinence. This model of community-based intensive care tends to demonstrate medical and legal effectiveness while being associated with greater care acceptability by patients. In France, very little data exists on the subject.

Médecins du Monde (NGO), in collaboration with the Public Prosecutor's department of Marseille, proposes the implementation of the AILSI strategy for people who homeless with severe psychiatric disorders and referred to referral procedures. The research unit EA 3279 - CEReSS is in charge of the independent evaluation of this innovative intervention.

This is an randomized coontrolled study, with two groups: AILSI group (intervention) and TAU group (usual services). A total of 169 patients will be included (80 in the AILSI group / 89 in the TAU group).

The main objective is to evaluate the effectiveness of the innovative program (AILSI) compared to usual services by assessing the duration of reincarceration at 18 months in each group, weighted by exposure time.

. Duration of inclusion: 39 months; Duration of follow-up: 18 months; Total duration of the study: 60 months.

Both quantitative and qualitative analyses will be conducted to address overall outcomes. Univariate and multivariate analyzes will be performed on the primary outcome as well as the secondary outcomes in order to highlight significant differences between the two groups and to identify predictive factors for improved effectiveness. The analysis will be conducted in accordance with Good Epidemiological Practices, and the final report will be written according to the CONSORT (Consolidated Standards of Reporting Trials) recommendations.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Being defered in referral procedures to the Public Prosecutor's department of Marseille
* Being homeless (ETHOS 1 to 8.3)
* Presenting a diagnosis of a severe psychiatric disorder as defined by DSM-IV-TR
* Having health coverage
* Having signed an informed consent to participate in the study
* Having declared to want to stay in the area at least 18 months after inclusion in the study.

Exclusion Criteria:

* Less than 18 years old;
* Do not have any criteria for ETHOS 1 to 8.3 classification
* Do not present a diagnosis of a severe psychiatric disorder as defined by DSM-IV-TR
* Presenting cognitive impairment that limits comprehension,
* Being under guardianship,
* Do not have health coverage
* Having refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
Duration of reincarceration, weighted by exposure time | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — AP-HM
Locations (1):
- Service Epidémiologie et Economie de la Santé - AP-HM, Marseille, France